CLINICAL TRIAL: NCT02303977
Title: Phase II Study of Abraxane and Gemicitabine in Patients With Advanced Adenocarcinoma Non-Small Cell Lung Cancer Progressing After First-Line Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 21514
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Patients With Stage IV or Recurrent Adenocarcinoma of the Lung
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: a prospective, single-arm, non-randomized, phase II trial designed to evaluate the efficacy of combination gemcitabine and albumin-bound paclitaxel for advanced adenocarcinoma non-small cell lung cancer progressing after first-line platinum-based chemotherapy.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine + Paciltaxel (Experimental): All patients were treated intravenously with albumin-bound paclitaxel at 100 mg/m2 plus gemcitabine at 1000 mg/m2 on days 1 and 8 of each three-week cycle.
  Interventions: Drug: Abraxane; Drug: Gemcitabine

INTERVENTIONS:
Drug: Abraxane
Drug: Gemcitabine

SUMMARY:
The main purpose of this study is to see how well the combination of Abraxane and gemcitabine works in people with advanced adenocarcinoma NSCLC who have already had treatment for their disease. Gemcitabine and Abraxane are FDA approved chemotherapies; however, the FDA has not approved this combination in the treatment of this specific type of cancer. Patients may continue to receive the study drugs until their disease gets worse or they have unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of adenocarcinoma non-small cell lung cancer
* Stage IV non-small cell lung cancer or recurrent disease which cannot be approached with curative intent.
* First-line treatment with a standard platinum doublet chemotherapy regimen (carboplatin or cisplatin at standard dosing plus one of the following drugs at standard dosing: paclitaxel, docetaxel, vinblastine, vinorelbine, pemetrexed, or etoposide). Patients who received platinum-based chemotherapy for localized lung cancer (either adjuvant chemotherapy following surgery or chemotherapy given in conjunction with definitive radiation) are eligible if their cancer has recurred within 6 months of platinum-based chemotherapy.
* Must have recovered from toxic effects of prior chemotherapy
* ECOG performance status of 0-1
* Life expectancy of at least 12 weeks
* Age 18 or greater
* Must have measurable disease defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded as > 20 mm with conventional techniques or > 10 mm with spiral CT scanning).
* Patients with prior malignancies are allowed, provided they have been treated with curative intent and have no evidence of active disease.
* Patients must be capable of giving informed consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
* Bilirubin < 1.5 mg/dL
* Patients must have adequate liver function: AST and ALT < 2.5 X upper limit of normal, alkaline phosphatase < 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
* Patients must have adequate bone marrow function: Platelets >100,000 cells/mm3, Hemoglobin > 9.0g/dL and ANC > 1,500 cells/mm3
* Patients must have adequate renal function: creatinine <1.5 mg/dL
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment
* Negative serum β-hCG pregnancy test at screening for patients of childbearing potential.
* Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE)

Exclusion Criteria:

* Patients with EGFR or EML4-ALK mutations
* ECOG performance status >1
* Patients previously treated with gemcitabine or Abraxane
* Uncontrolled intercurrent illness including, but not limited to: uncontrolled ongoing infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV or Hepatitis C
* Untreated central nervous system metastases. Patients are eligible if they are clinically stable, off all steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, stereotactic radio surgery) ending at least 2 weeks prior to enrollment, or after surgical resection performed at least 2 weeks prior to enrollment.
* Concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemo-embolization, targeted therapy, or an investigational agent
* Pregnant or breast-feeding patients, as chemotherapy is thought to present substantial risk to the fetus/infant. Men and women of reproductive potential may not participate in this study unless they have agreed to use an effective contraceptive method while in this study. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients must agree to continue contraception for 3 months from the date of the last study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ciunci, MD, Principal Investigator — Abramson Cancer Center

REFERENCES:
- [Derived] Ciunci CA, Reibel JB, Evans TL, Mick R, Bauml JM, Aggarwal C, Marmarelis ME, Singh AP, D'Avella C, Cohen RB, Langer CJ. Phase II Trial of Combination Nab-paclitaxel and Gemcitabine in Non-squamous Non-small Cell Lung Cancer After Progression on Platinum and Pemetrexed. Clin Lung Cancer. 2022 Jun;23(4):e310-e316. doi: 10.1016/j.cllc.2022.02.004. Epub 2022 Mar 14. PMID 35393247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine + Paciltaxel
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Paciltaxel
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 66 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The percentage of patients with a Partial Response or Complete Response recorded from the start of the treatment until disease progression/recurrence by RECIST 1.1 criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Averaging about 16 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine + Paciltaxel
Number analyzed (Participants) | 37
percentage of participants | 13.5 [2.5 to 24.5]

2. Secondary Outcome: Progression-free Survival
Description: Measures the length of time from the first day of therapy until Progressive Disease, death from any cause, or last patient contact. Disease Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Averaging about 16 weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine + Paciltaxel
Number analyzed (Participants) | 37
Months | 2.6 [1.4 to 3.8]

3. Secondary Outcome: Overall Survival
Description: Length of time from the first day of therapy to death from any cause or last patient contact
Time Frame: Averaging about 47 weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine + Paciltaxel
Number analyzed (Participants) | 37
Months | 6.2 [4.2 to 8.2]

4. Secondary Outcome: Disease Control Rate
Description: The percentage of patients with a Partial Response, a Complete Response, or Stable Disease during the study. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: The duration of study treatment, averaging about 16 weeks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Gemcitabine + Paciltaxel: All patients were treated intravenously with albumin-bound paclitaxel at 100 mg/m2 plus gemcitabine at 1000 mg/m2 on days 1 and 8 of each three-week cycle.
  Abraxane
  Gemcitabine
Arm/Group | Gemcitabine + Paciltaxel
Number analyzed (Participants) | 37
Percentage of participants | 59.5 [43.5 to 75.5]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of the initiation of study treatment, until 30 days after the end of study treatment, for an average of about 20 weeks. All-Cause Mortality was assessed from the time of study initiation until the death of the subject by any cause, up to approximately 47 weeks.
Arm/Group | Gemcitabine + Paciltaxel
All-Cause Mortality (participants affected / at risk) | 36/37
Serious Adverse Events (participants affected / at risk) | 22/37
Other Adverse Events (participants affected / at risk) | 34/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Paciltaxel (N=37)
Vomitting (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lung Infection (Infections and infestations) | 5 (5)
Myelitis (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
thromboembolic event (Vascular disorders) | 7 (7)
anemia (Blood and lymphatic system disorders) | 3 (3)
ANC Decreased (Infections and infestations) | 4 (4)
Failure to thrive (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
WBC decreased (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 2 (2)
Tumor invasion of left brachial plexus (Nervous system disorders) | 1 (1)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Paciltaxel (N=37)
Fatigue (General disorders) | 19
Anemia (Blood and lymphatic system disorders) | 17
Nausea (Gastrointestinal disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 11
Neutrophil count decreased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 9
Diarrhea (Gastrointestinal disorders) | 7
Fever (General disorders) | 7
Vomitting (Gastrointestinal disorders) | 7
Platelet count decreased (Investigations) | 6
ALT increased (Investigations) | 5
Neuropathy (Nervous system disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
White blood cell decreased (Blood and lymphatic system disorders) | 5
AST Increased (Investigations) | 4
Constipation (Gastrointestinal disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT02303977/Prot_SAP_000.pdf